CLINICAL TRIAL: NCT00814255
Title: Novel Therapies for Resistant Focal Segmental Glomerulosclerosis
Brief Title: Novel Therapies for Resistant FSGS (FONTII): Phase II Clinical Trial
Acronym: FONTII
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: University of Michigan (Other); The Cleveland Clinic (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DK70341FII; R33DK070341 (NIH)
Record Dates: First submitted 2008-12-22; First posted 2008-12-24 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Focal Segmental Glomerulosclerosis
Keywords: Primary FSGS; Steroid Resistant; Rosiglitazone; Adalimumab; Resistant primary FSGS; GALACTOSE
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental | interventions — Adalimumab; Lisinopril; Losartan; Atorvastatin; Galactose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 2 (Experimental): Conservative medical therapy plus adalimumab
  Interventions: Drug: Adalimumab
- 1 (Active Comparator): Conservative medical therapy (lisinopril, losartan, atorvastatin)
  Interventions: Drug: Lisinopril, losartan, and atorvastatin
- conservative medical therapy plus galactose (Experimental): drug: galactose 0.2 g /kg/dose (maximum dose 15g) po BID
  Interventions: Drug: galactose

INTERVENTIONS:
Drug: Adalimumab — Adalimumab 24 mg/m^2 (maximum dose 40 mg) sc q 14 days
  Arms: 2
Drug: Lisinopril, losartan, and atorvastatin — Lisinopril PO 10-20 mg per day Losartan PO 25-50 mg per day Atorvastatin PO 10-20 mg per day
  Arms: 1
Drug: galactose — galactose 0.2 g/kg/dose (maximum dose 15 g)po BID
  Arms: conservative medical therapy plus galactose

SUMMARY:
This project will test whether adalimumab,and/or galactose can safely reduce proteinuria (abnormal amounts of protein in the urine) and protect kidney function better than standard treatment for patients with focal segmental glomerulosclerosis (FSGS).

DETAILED DESCRIPTION:
SPECIFIC AIMS A significant percentage of patients with primary FSGS are resistant to corticosteroids and other immunosuppressive medications. In view of the rising incidence of this disease and the grim prognosis for patients with resistant disease, it is imperative that new therapeutic approaches be evaluated in an efficient and systematic manner. This will enable accurate assessment of the risk-benefit ratio of novel therapies and guide the design of future Phase III randomized clinical trials.

Specific Aim #1: To evaluate two novel therapies for resistant FSGS -- anti-TNF-α antibody and galactose -- against standard therapy

Specific Aim #2: To identify one or more novel agents as candidates for future study in a Phase III randomized clinical trial

OVERALL STUDY DESIGN Screening/Run-In: There is no formal run-in period in the phase II trial because patients with resistant FSGS who will be eligible for this study often have unstable kidney function and are prone to sudden decline in glomerular filtration rate (GFR). An effort will be made to achieve randomization within 2 weeks of the screening visit.

In order to achieve a comparable baseline assessment prior to initiation of one of the novel therapies, the patients must be off all immunosuppressive medications for 30 days. In addition, patients will be placed on the maximal tolerated doses of an angiotensin-converting enzyme inhibitor (ACEI), an angiotensin receptor blocker (ARB), and a lipid-lowering drug defined above based upon measurements of blood pressure, serum K+, creatinine, and cholesterol concentrations. Patients will have to be on stable doses of the ACEI/ARB treatment for a minimum of 2 weeks prior to randomization into the FONT Phase II study to insure that the initiation of novel therapy does not coincide with a hemodynamically induced change in proteinuria. In order to implement this part of conservative medical therapy, a 2-12 week Screening/Run-In period will precede randomization. Rescreening will be necessary if patients are not randomized to one of the three treatment arms within 12 weeks of the initial screening assessment.

Duration of novel therapy: Novel therapies will be administered for 6 months before assessing efficacy, i.e., >50% reduction in proteinuria. Although the novel therapies target renal fibrosis, it is anticipated that this period of treatment will be sufficient to document a beneficial effect on proteinuria.

Screening/Run-In: There is no formal run-in period in the phase II trial because patients with resistant FSGS who will be eligible for this study often have unstable kidney function and are prone to sudden decline in GFR. An effort will be made to achieve randomization within 2 weeks of the screening visit.

Frequency of visits: Patients will be evaluated after 0, 2, 8, 16, and 26 weeks of treatment with the novel therapy or conservative medical therapy alone. Thus, there will be a total of 6 visits during the treatment period. A follow-up evaluation will be performed at 1 month, 3 months, and 6 months after discontinuation of the novel therapy, and then every 6 months until the end of the funding period.

Baseline studies

1. Interval History and physical examination
2. Urine protein and creatinine excretion Proteinuria (Up/c) will be expressed as the protein: creatinine ratio (mg: mg) in an early morning specimen.
3. Serum creatinine and calculated GFR, glucose, albumin, pregnancy test
4. A urine, plasma, serum and DNA sample will be collected for storage in the NIDDK FSGS-CT Biorepository. A request will be made to store any residual renal tissue collected for clinical indications during the FONT trial in the NIDDK Biorepository.

Follow-up assessment: Week 2, 8, and 16 Visits

1. Interval history, physical examination, assessment of adverse events
2. First morning urine protein excretion
3. Laboratory analysis as charted below. Urine pregnancy test at 8 and 16 week visit

Final Outcome Visit (Week 26)

1. History and physical examination
2. Morning urine protein and creatinine excretion x 2 (The value will represent the average of two samples collected during the week before the visit.)
3. Serum creatinine and calculated GFR, Serum Na+, K+, HCO3, Cl-, glucose, CPK
4. Blood urea nitrogen (BUN), albumin, cholesterol, aspartate transaminase (AST), alanine transaminase (ALT), alkaline phosphatase, complete blood count (CBC), antinuclear antibodies (ANA), C3 levels, pregnancy test
5. Urine, serum and plasma for biorepository
6. TSQM patient questionnaire

Preliminary safety, patient tolerance, and pharmacokinetic (PK) data for the two novel therapies, rosiglitazone and adalimumab, that will be used in the Phase II trial were generated through the successful performance of a Phase I study.

In the phase I study, a total of 21 patients were enrolled. 11 were assigned to receive rosiglitazone, and 10 were assigned to receive adalimumab. The patients were evenly divided by gender and pubertal stage. All patients had a GFR >50 mL/min/1.73 m2.

There were no serious adverse events necessitating the withdrawal of study drug.

Rosiglitazone was stopped in one child due to a questionable allergy. The patients tolerated the experimental medications adequately based on the results of the Treatment Satisfaction Questionnaire for Medication (TSQM) which was administered at week 16.

The PK analyses indicated that the rosiglitazone dose needs to be increased to account for increased clearance and reduced area under the curve in patients with resistant FSGS and nephrotic range proteinuria. For adalumimab, clearance was also enhanced especially after receiving multiple doses. However, these results of the adalimumab PK analyses indicate that no dose adjustment was required.

The PK data for each drug were presented in abstract form at the annual meeting of the American Society of Nephrology and a manuscript summarizing the complete findings in patients treated with rosiglitazone has been submitted for publication.

This Phase II will again rely on the considerable investment of time and resources on the part of the study investigators and the NIH/NIDDK gained through the FSGS-CT (UO1-DK-63455) and the Phase I portion of the FONT study (DK70341). Schneider Children's Hospital (SCH) and University of North Carolina-Chapel Hill (UNC) resources including the GCRCs that were utilized in the R21phase of them study will be available for the R33 portion of the FONT project.

ELIGIBILITY:
Inclusion Criteria:

* Primary FSGS confirmed by renal biopsy OR documentation of a genetic mutation in a podocyte protein associated with the disease
* Failure to respond to prior therapy at least one of the following immunosuppressive medications -- cyclosporine, tacrolimus, mycophenolate mofetil, sirolimus - or other agents prescribed to lower proteinuria
* Age 1-65 years at onset of proteinuria
* Age 1-65 years at time of randomization
* Estimated GFR ≥40 mL/min/1.73 m2 using Schwartz (age <18 yr) or Cockroft-Gault (age <18 yr) formula at screening and ≥30 mL/min/1.73 m2 at the end of the Run-In Period and at the time of randomization
* Up/c > 1.0 g/g creatinine on first morning void
* Steroid resistance defined as failure to achieve sustained Up/c < 1.0 following a standard course of prednisone/prednisolone/methylprednisolone prescribed for FSGS therapy, OR contraindication/anticipated intolerance to steroid therapy defined as severe obesity, documented decreased bone density, family history of diabetes, or a psychiatric disorder.
* Willingness to follow the protocol, including medications, baseline and follow-up visits, and procedures.

Exclusion Criteria:

* Lactation, pregnancy, or refusal of birth control in women of child bearing potential
* Participation in another therapeutic trial involving protocol mandated administration of a immunosuppressive medication concurrently or 30 days prior to randomization
* Active/serious infection (including, but not limited to Hepatitis B or C, HIV)
* History of malignancy
* Abnormality in age appropriate cancer screening in accord with ACS 2003 guidelines (appendix 17.6)
* Patients with uncontrolled blood pressure > 140/90 or > 95th percentile for age/height at the end of the run in period
* Diabetes mellitus Type I or II
* Organ transplantation
* Congestive heart failure
* History of prior myocardial infarction
* SLE or multiple sclerosis
* Hepatic disease, defined as serum ALT/AST levels more than 2.5x the upper limit of normal
* Hematocrit <27%
* Immunosuppressive therapy with cyclosporine, tacrolimus, mycophenolate mofetil, azathioprine, or rapamycin in the 30 days prior or Rituximab in the 90 days prior to randomization
* Prior treatment with the study medications, rosiglitazone or adalimumab
* Allergy to one of the study medications, i.e., rosiglitazone, adalimumab, lisinopril, losartan or atorvastatin

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-12; Primary Completion 2013-06 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Howard Trachtman, MD, Principal Investigator — NYU Langone Medical Center; Debbie Gipson, MD, Principal Investigator — University of Michigan; Jennifer Gassman, PhD, Principal Investigator — The Cleveland Clinic
Locations (18):
- United States (17):
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - University of Kansas, Kansas City, Kansas
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - NYU Langone Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Doernbecher Children's Hospital, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Tech University, El Paso, Texas
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
will comply with NIDDK guidelines

REFERENCES:
- [Result] Joy MS, Gipson DS, Dike M, Powell L, Thompson A, Vento S, Eddy A, Fogo AB, Kopp JB, Cattran D, Trachtman H. Phase I trial of rosiglitazone in FSGS: I. Report of the FONT Study Group. Clin J Am Soc Nephrol. 2009 Jan;4(1):39-47. doi: 10.2215/CJN.02310508. Epub 2008 Dec 10. PMID 19073787
- [Result] Trachtman H, Vento S, Herreshoff E, Radeva M, Gassman J, Stein DT, Savin VJ, Sharma M, Reiser J, Wei C, Somers M, Srivastava T, Gipson DS. Efficacy of galactose and adalimumab in patients with resistant focal segmental glomerulosclerosis: report of the font clinical trial group. BMC Nephrol. 2015 Jul 22;16:111. doi: 10.1186/s12882-015-0094-5. PMID 26198842
- [Derived] Liu ID, Willis NS, Craig JC, Hodson EM. Interventions for idiopathic steroid-resistant nephrotic syndrome in children. Cochrane Database Syst Rev. 2025 May 8;5(5):CD003594. doi: 10.1002/14651858.CD003594.pub7. PMID 40337980
- [Derived] Hodson EM, Sinha A, Cooper TE. Interventions for focal segmental glomerulosclerosis in adults. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD003233. doi: 10.1002/14651858.CD003233.pub3. PMID 35224732
- [Derived] Trachtman H, Vento S, Gipson D, Wickman L, Gassman J, Joy M, Savin V, Somers M, Pinsk M, Greene T. Novel therapies for resistant focal segmental glomerulosclerosis (FONT) phase II clinical trial: study design. BMC Nephrol. 2011 Feb 10;12:8. doi: 10.1186/1471-2369-12-8. PMID 21310077
- [Derived] Joy MS, Gipson DS, Powell L, MacHardy J, Jennette JC, Vento S, Pan C, Savin V, Eddy A, Fogo AB, Kopp JB, Cattran D, Trachtman H. Phase 1 trial of adalimumab in Focal Segmental Glomerulosclerosis (FSGS): II. Report of the FONT (Novel Therapies for Resistant FSGS) study group. Am J Kidney Dis. 2010 Jan;55(1):50-60. doi: 10.1053/j.ajkd.2009.08.019. Epub 2009 Nov 22. PMID 19932542

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 32 patients consented however 8 were not assigned to treatment because they failed to meet eligibility at the end of the screening
  1 patient was assigned to rosiglitazone and was not included in the analysis.
Groups:
- Conservative Medical Therapy Plus Adalimumab: Conservative medical therapy plus adalimumab
  Adalimumab: Adalimumab 24 mg/m2 (maximum dose 40 mg) sc q 14 days
- Conservative Medical Therapy (Lisinopril, Losartan, Atorvastat: Conservative medical therapy (lisinopril, losartan, atorvastatin)
  Lisinopril, losartan, and atorvastatin: Lisinopril PO 10-20 mg per day Losartan PO 25-50 mg per day Atorvastatin PO 10-20 mg per day
- Conservative Medical Therapy Plus Galactose: drug: galactose 0.2 g /kg/dose (maximum dose 15g) po BID
  galactose: galactose 0.2 g/kg/dose (maximum dose 15 g)po BID
  NOTE: This study arm was originally to receive rosiglitazone. One participant was assigned to this study arm prior to the therapy being changed to galactose.
Period: Overall Study
Arm/Group | Conservative Medical Therapy Plus Adalimumab | Conservative Medical Therapy (Lisinopril, Losartan, Atorvastat | Conservative Medical Therapy Plus Galactose
Started | 8 | 7 | 8
Completed | 7 | 7 | 7
Not Completed | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Conservative Medical Therapy: Conservative medical therapy (lisinopril, losartan, atorvastatin)
  Lisinopril, losartan, and atorvastatin: Lisinopril PO 10-20 mg per day Losartan PO 25-50 mg per day Atorvastatin PO 10-20 mg per day
- Total: Total of all reporting groups
Arm/Group | Conservative Medical Therapy Plus Adalimumab | Conservative Medical Therapy | Conservative Medical Therapy Plus Galactose | Total
Number analyzed (Participants) | 7 | 7 | 7 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 5 | 4 | 14
  Between 18 and 65 years | 2 | 2 | 3 | 7
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 21.9 [7.2 to 36.7] | 15.6 [3.8 to 34.1] | 15.8 [13 to 21] | 17.8 [3.8 to 36.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 4 | 12
  Male | 3 | 3 | 3 | 9
Race/Ethnicity, Customized [Number; unit: participants]
  white | 3 | 7 | 2 | 12
  hispanic | 2 | 0 | 3 | 5
  African American | 2 | 0 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 7 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Reduction in Proteinuria at 6 Months by > 50% of the Value at Screening AND Stable GFR Defined as Greater Than 75 ml/Min/1.73m2 in Those With an Initial Value Above 90 OR Within 25% of Baseline for Remaining Patients
Description: Number of participants with a reduction in proteinuria at 6 months by > 50% of the value at screening AND stable GFR defined as greater than 75 ml/min/1.73m2 in those with an initial value above 90 OR within 25% of baseline for remaining patients.
Time Frame: baseline and 6 months
Population: One participant was assigned to the rosiglitazone arm before the drug was replaced with the galactose arm. This participant was not included in the analysis.
Measure: Number; unit: participants
Groups:
- Conservative Medical Therapy Plus Adalimumab: Conservative medical therapy plus adalimumab
  Adalimumab: Adalimumab 24 mg/m2 (maximum dose 40 mg) sc q 14 days 0 out of 7
- Conservative Medical Therapy (Lisinopril, Losartan, Atorvastat: Conservative medical therapy (lisinopril, losartan, atorvastatin)
  Lisinopril, losartan, and atorvastatin: Lisinopril PO 10-20 mg per day Losartan PO 25-50 mg per day Atorvastatin PO 10-20 mg per day 2 out of 7
- Conservative Medical Therapy Plus Galactose: drug: galactose 0.2 g /kg/dose (maximum dose 15g) po BID
  galactose: galactose 0.2 g/kg/dose (maximum dose 15 g)po BID 2 out of 7
Arm/Group | Conservative Medical Therapy Plus Adalimumab | Conservative Medical Therapy (Lisinopril, Losartan, Atorvastat | Conservative Medical Therapy Plus Galactose
Number analyzed (Participants) | 7 | 7 | 7
participants | 0 | 2 | 2

2. Secondary Outcome: Patient Satisfaction Score Using the Treatment Satisfaction Questionnaire for Medication (TSQM Questionnaire)
Description: Patient Satisfaction Score Using the Treatment Satisfaction Questionnaire for Medication (TSQM Questionnaire)
Time Frame: Baseline and 6 months
Population: No data were collected.
Arm/Group | Conservative Medical Therapy Plus Adalimumab | Conservative Medical Therapy (Lisinopril, Losartan, Atorvastat | Conservative Medical Therapy Plus Galactose
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Adverse Events
Time Frame: Up to 7 months
Measure: Number; unit: participants
Arm/Group | Conservative Medical Therapy Plus Adalimumab | Conservative Medical Therapy (Lisinopril, Losartan, Atorvastat | Conservative Medical Therapy Plus Galactose
Number analyzed (Participants) | 7 | 7 | 7
participants | 7 | 7 | 7

4. Secondary Outcome: Percent Change in Proteinuria
Time Frame: Baseline and 6 months
Population: No data were collected.
Arm/Group | Conservative Medical Therapy Plus Adalimumab | Conservative Medical Therapy (Lisinopril, Losartan, Atorvastat | Conservative Medical Therapy Plus Galactose
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Percent Change in or Time to Doubling of Serum Creatinine
Time Frame: Baseline and 6 months
Population: No data were collected.
Arm/Group | Conservative Medical Therapy Plus Adalimumab | Conservative Medical Therapy (Lisinopril, Losartan, Atorvastat | Conservative Medical Therapy Plus Galactose
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 month treatment period and 6 month follow up period
Description: Data collected based on patient reports and a review of laboratory data. Adverse events were classified by MeDRA 10.0
Arm/Group | Conservative Medical Therapy Plus Adalimumab | Conservative Medical Therapy (Lisinopril, Losartan, Atorvastat | Conservative Medical Therapy Plus Galactose
Serious Adverse Events (participants affected / at risk) | 3/7 | 1/7 | 1/7
Other Adverse Events (participants affected / at risk) | 7/7 | 7/7 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conservative Medical Therapy Plus Adalimumab (N=7) | Conservative Medical Therapy (Lisinopril, Losartan, Atorvastat (N=7) | Conservative Medical Therapy Plus Galactose (N=7)
hospitalization (General disorders) | 3 (32) | 1 (9) | 1 (1) — Hospitalization 5 patients
Pregnancy (General disorders) | 1 (1) | 0 (0) | 1 (1) — Pregnancy
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conservative Medical Therapy Plus Adalimumab (N=7) | Conservative Medical Therapy (Lisinopril, Losartan, Atorvastat (N=7) | Conservative Medical Therapy Plus Galactose (N=7)
Edema (General disorders) | 6 (100) | 6 (23) | 5 (57) — Edema
Infection (Infections and infestations) | 5 (49) | 4 (10) | 5 (20) — Infection

LIMITATIONS AND CAVEATS:
1. Limited sample size
2. Extended enrollment period
3. Replacement of rosiglitazone with galactose after start of trial

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No